CLINICAL TRIAL: NCT02173743
Title: Calcific Tendinitis of the Rotator Cuff: a Randomized Controlled Trial to the Effects of the Adjuvant Application of Platelet-rich Plasma After Needle Aspiration of Calcific Deposits
Brief Title: Platelet-rich Plasma in Calcific Tendinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopedisch Centrum Oost Nederland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL47402.044.13; ABR 47402 (Other: Medical Ethical Committee Twente)
Record Dates: First submitted 2014-06-19; First posted 2014-06-25 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Calcific Tendinitis
Keywords: plasma, calcific tendinitis, rotator cuff, PRP

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRP group (Experimental): PRP during barbotage
  Interventions: Other: PRP
- Control group (Other): Regular barbotage
  Interventions: Other: Control

INTERVENTIONS:
Other: PRP — platelet enriched autologous blood plasma
  Arms: PRP group
Other: Control — Regular barbotage/care as usual
  Arms: Control group

SUMMARY:
Needle aspiration of calcific deposits (NACD ) is the treatment of choice for calcific tendinitis which does not respond to conservative treatment. NACD is effective in approximately 70% of the patients.When NACD is not effective, surgery is often the only treatment that remains.Surgery, however, is discouraged by th e Dutch guidelines for diagnosing and treating patients with subacromial pain syndrome.Therefore,both patients and the doctors treating those patients will benefit from a more effective minimal invasive treatment for calcific tendinitis.Injection of platelet-rich plasma (PRP) might, considering its positive effect on tissue repair, be a possible solution here.Previous research investigating the effects of PRP on other tendinopathies did, however, show controversial results. The aim of this double-blind randomized controlled trial is to investigate the effect of the adjuvant application of PRP after NACD on pain reduction ,recovery of shoulder function, tendon recovery,resorption of calcific deposits, the percentage of patients with persistent complaints and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 yrs
* clinical manifestions of tendinitis calcarea (pain, stifness, lock sensations, muscle atrophy)
* persistent pain sympoms >6 months
* standardized AP x-ray shows calcific deposit of > 5mm & morphologic Type I & II deposits (classification of Gärtner en Simons)
* ineffective intervention > 2 types of conservative treatment (among which are non-steroidal anti-inflammatory drugs, physiotherapy, local anesthesia injection and/or corticosteroids, extracorporele shock wave therapy)
* indication and referral for barbotage by orthopeadic surgeon

Exclusion Criteria:

* age > 55 years
* morphological type III deposits according to classification of Gärtner and Simons) (as indicated by standardized x-ray AP)
* bigliani type III acromion, and acromial spur of acromioclavicular osteovyt
* previous (ineffective) barbotage
* the existence of other shoulder related injuries next to calcific tendinitis (full-thickness rupture of the rotator cuff, adhesive capsulitis (frozen shoulder), arthrosis of the glenohumeral- or acromioclavicalar joint
* shoulder joint instability
* shoulder injury due to trauma or previous shoulder surgeries
* other types of disorders that could negatively influence the outcomes (rheumatic arthritis. cervical spine disorders, neurological upper extremity disorders, diabetes mellitus, infections, blood disorders, malignity, pregnancy)
* known allergic responses to one of the medications applied in the current study (lidocaine, bupivacaine, kenacort)
* usage of anti-coagulants other than ascal of plavix

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-07; Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) pain | 6 months post barbotage
  Score to assess the amount of pain

SECONDARY OUTCOMES:
Constant-Murley Score (CMS) | 6 weeks, 3 - 6- 12- 25 months post barbatoge
  To assess shoulder function
Quality of Life (EQ-5D) | 6 weeks, 3- 6- 12- 24 months post barbotage
  score to assess the quality of life

OTHER OUTCOMES:
Tendon recovery | 6 weeks, 3-6-12-24 months post barbotage
  to visualize tendon recovery by ultrasound
calcifications | baseline, 3 + 12 months post barbotage
  size of calcifications (X-ray)
plated plasma analysis | baseline
  trombocytes analysis of PRP blood

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Ooms, PhD, Study Director — OCON; Rianne Huis in 't Veld, PhD, Study Director — OCON; Bart Oudelaar, MSc, Principal Investigator — OCON
Locations (1):
- Orthopedisch Centrum Oost Nederland/ZGT, Hengelo, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Oudelaar BW, Huis In 't Veld R, Ooms EM, Schepers-Bok R, Nelissen RGHH, Vochteloo AJH. Efficacy of Adjuvant Application of Platelet-Rich Plasma After Needle Aspiration of Calcific Deposits for the Treatment of Rotator Cuff Calcific Tendinitis: A Double-Blinded, Randomized Controlled Trial With 2-Year Follow-up. Am J Sports Med. 2021 Mar;49(4):873-882. doi: 10.1177/0363546520987579. Epub 2021 Feb 10. PMID 33566629
- See also: hospital's url — http://www.ocon.nl